CLINICAL TRIAL: NCT02138253
Title: A Multicenter, Double-Blind, Randomized Trial of IDN-6556 in Subjects Who Had Hepatitis C Virus (HCV) Reinfection and Liver Fibrosis Following Orthotopic Liver Transplantation for Chronic HCV Infection and Who Subsequently Achieved a Sustained Virologic Response Following Anti-HCV Therapy
Brief Title: A Trial of IDN-6556 in Post Orthotopic Liver Transplant for Chronic HCV
Acronym: POLT-HCV-SVR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Conatus Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IDN-6556-07
Record Dates: First submitted 2014-05-12; First posted 2014-05-14 (Estimated); Results first posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-11

CONDITIONS: Liver Fibrosis; Hepatic Fibrosis; Liver Cirrhosis; Hepatic Cirrhosis
Keywords: liver transplant; hepatitis C; liver fibrosis; hepatic fibrosis; liver cirrhosis; hepatic cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis C | interventions — 3-(2-(2-tert-butylphenylaminooxalyl)aminopropionylamino)-4-oxo-5-(2,3,5,6-tetrafluorophenoxy)pentanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IDN-6556 (Experimental): IDN-6556 25 mg BID
  Interventions: Drug: IDN-6556
- Placebo (Placebo Comparator): Placebo BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IDN-6556
  Other Names: emricasan; PF-03491390
  Arms: IDN-6556
Drug: Placebo — Placebo control
  Arms: Placebo

SUMMARY:
This is a double-blind, multicenter study involving patients with chronic HCV infection who had a liver transplantation; developed HCV-related liver fibrosis and/or incomplete cirrhosis; achieved a sustained virologic response (SVR) following anti-HCV therapy; but still have fibrosis and/or incomplete cirrhosis on liver biopsy to see if treatment with IDN-6556 is better than placebo in reversing or stopping the progression of the damage to the new liver caused by HCV.

DETAILED DESCRIPTION:
There are data to suggest that with eradication of the HCV virus, improvements in liver fibrosis can be seen in the post-transplant population. However, amelioration of inflammatory activity, and deceleration of fibrosis progression is a gradual process over the course of many years. This placebo-controlled study is designed to evaluate the effects of IDN-6556, compared to placebo, on markers of apoptosis and inflammation, and liver histology.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of minimum adult legal age (according to local laws for signing the informed consent document), able to provide written informed consent, and able to understand and willing to comply with the requirements of the study
* History of orthotopic liver transplantation for HCV-induced liver disease
* Diagnosis of HCV infection (HCV-RNA detectable in serum) and liver fibrosis and/or incomplete cirrhosis status post liver transplantation, and achieved a sustained virologic response (SVR) with anti-viral HCV treatment within 18 months of Day 1
* Liver fibrosis on liver histology as read by central histopathologist of Ishak F2 to F6 within three months of Day 1 (Up to 15 subjects with an Ishak score of F6 can be enrolled)
* Willingness to utilize two reliable forms of contraception (for both males and females of childbearing potential) from Screening to one month after the last dose of study drug

Exclusion Criteria:

* Known infection with hepatitis B virus (HBV) and/or human immunodeficiency virus (HIV)
* History of renal transplant and/or severe renal impairment defined as eGFR (estimated glomerular filtration rate) of less than 30 mL/min/1.73 m2
* Evidence of tumor burden >Milan criteria, or evidence of micro- or macrovascular invasion in explanted liver
* Hepatocellular carcinoma (HCC) at entry into the study
* Concurrent sirolimus (rapamycin) use
* History or presence of clinically concerning cardiac arrhythmias, or prolongation of Screening (pre-treatment) QT or QTc interval of > 480 milliseconds (msec)
* Subjects with diagnosed or suspected systemic lupus erythematosus (SLE) and/or rheumatoid arthritis (RA)
* If female: known pregnancy, positive urine or serum pregnancy test, or lactating/breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-05; Primary Completion 2018-02-15 (Actual); Study Completion 2018-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hagerty, MD, Study Chair — Conatus Pharmaceuticals Inc.
Locations (35):
- United States (35):
  - Southern California Research Center, Coronado, California
  - Scripps Clinic, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - UCLA Pfleger Liver Institute, Los Angeles, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Johns Hopkins Sibley Memorial Hospital, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - Tulane Health Science Center, New Orleans, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - John Hopkins Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henery Ford Health System, Detroit, Michigan
  - Saint Louis University, St Louis, Missouri
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Columbia University Medical Center, New York, New York
  - University of Cincinnati Physicians Company, Cincinnati, Ohio
  - University of Pennsylvania Milton Hershey Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Baylor All Saints Medical Center, Fort Worth, Texas
  - Liver Associates of Texas, PA, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - VAMC/Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Bon Secours Mary Immaculate Hospital, Newport News, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, Richmond, Virginia
  - McGuire DVAMC, Richmond, Virginia
  - University of Washington Harborview Medical Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 20 of 35 US sites that obtained IRB approval. First subject randomized Sep 2014, last subject last visit was 15 Feb 2018.
  A total of 114 subjects were screened, 64 subjects randomized with 41 subjects randomized to emricasan and 23 subjects randomized to placebo. Thirteen subjects discontinued the study.
Groups:
- IDN-6556: IDN-6556 25 mg BID
  IDN-6556
Period: Overall Study
Arm/Group | IDN-6556 | Placebo
Started | 41 | 23
Completed | 32 | 19
Not Completed | 9 | 4
Not completed — Adverse Event | 3 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Non compliance | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who underwent orthotopic liver transplantation for chronic HCV, developed HCV-related liver fibrosis or cirrhosis, achieved a SVR with anti-viral treatment and had demonstrable fibrosis or cirrhosis on liver histology were enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDN-6556 | Placebo | Total
Number analyzed (Participants) | 41 | 23 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 17 | 46
  >=65 years | 12 | 6 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 32 | 18 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 31 | 17 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 2 | 9
  White | 30 | 20 | 50
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 41 | 23 | 64
Baseline Ishak Fibrosis Score [Number; unit: participants] — Ishak Fibrosis Score is a standard measure to classify the severity of fibrosis in patients. A score of 0 indicates no evidence of fibrosis and a score of 6 indicates the most severe evidence of fibrosis (i.e., cirrhosis).
  participants
    Baseline Ishak Fibrosis Score F2 | 9 | 6 | 15
    Baseline Ishak Fibrosis Score F3 | 20 | 7 | 27
    Baseline Ishak Fibrosis Score F4 | 5 | 5 | 10
    Baseline Ishak Fibrosis Score F5 | 2 | 2 | 4
    Baseline Ishak Fibrosis Score F6 | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With At Least a One Stage Reduction From Baseline in Ishak Fibrosis Score
Description: At least a one stage reduction from baseline in Ishak Fibrosis Stage. Score F0 No fibrosis F1 Fibrous expansion of some portal areas, with or without short fibrous septa F2 Fibrous expansion of most portal areas, with or without short fibrous septa F3 Fibrous expansion of most portal areas, with occasional portal to portal bridging F4 Fibrous expansion of portal areas, with marked bridging (portal to portal as well as portal to central) F5 Marked bridging (portal to portal and/or portal to central) with occasional nodules (incomplete cirrhosis) F6 Cirrhosis probable or definite
  Since the primary analysis used multiple imputation methodology, the numerator and denominator varied across 20 imputations.
Time Frame: 24 months
Population: The Full Analysis Set (FAS) consisted of all randomized subjects who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 41 | 23
participants | 25 | 14
Statistical Analysis 1: Comparison: IDN-6556 vs Placebo; All screening and post-baseline biopsy data collected were used in the primary analysis, irrespective of the defined protocol visit window. Classification of the Ishak fibrosis score was summarized descriptively by treatment group at baseline, Month 12, and Month 24. Response at Months 12 and 24 were summarized descriptively by treatment group, along with exact (Clopper-Pearson) 95% confidence intervals (CIs). The risk difference between groups was also was provided with its 95% CI; Test type: Superiority — For the primary efficacy analysis based on the Month 24 biopsy, subjects with a missing Month 24 biopsy had their Ishak fibrosis score imputed. Imputation of missing Ishak fibrosis scores was conducted using multiple imputation (MI). Results were imputed based on age, gender, baseline Ishak fibrosis score, and the Month 12 Ishak fibrosis score; p = 0.73, Cochran-Mantel-Haenszel — Stratified by baseline Ishak Fibrosis Score strata (F2, F3+F4+F5, and F6); Risk Difference (RD) = 2.9, 95% CI 2-sided [-20.5 to 26.4]

2. Secondary Outcome: Number of Participants With At Least a One Stage Reduction From Baseline in Ishak Fibrosis Score (Observed Cases Only)
Description: At least a one stage reduction from baseline in Ishak Fibrosis Stage. Score F0 No fibrosis F1 Fibrous expansion of some portal areas, with or without short fibrous septa F2 Fibrous expansion of most portal areas, with or without short fibrous septa F3 Fibrous expansion of most portal areas, with occasional portal to portal bridging F4 Fibrous expansion of portal areas, with marked bridging (portal to portal as well as portal to central) F5 Marked bridging (portal to portal and/or portal to central) with occasional nodules (incomplete cirrhosis) F6 Cirrhosis probable or definite
Time Frame: 24 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 32 | 19
Participants | 25 | 14
Statistical Analysis 1: Comparison: IDN-6556 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.658, Cochran-Mantel-Haenszel; Risk Difference (RD) = 4.4, 95% CI 2-sided [-20.0 to 28.9]

3. Secondary Outcome: Number of Participants With At Least a One Stage Reduction From Baseline in Ishak Fibrosis Score
Description: as for outcome 2
Time Frame: 12 months
Population: Full analysis set, the # of subject analyzed included subjects with an observed Ishak Fibrosis Score at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 35 | 20
Participants | 27 | 17
Statistical Analysis 1: Comparison: IDN-6556 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.421, Cochran-Mantel-Haenszel; Risk Difference (RD) = -7.9, 95% CI 2-sided [-28.8 to 13.1]

4. Secondary Outcome: Alanine Aminotransferase (ALT) - Change From Baseline
Description: Liver function laboratory parameter
Time Frame: Baseline and 24 months
Population: Full analysis set, the # of subject analyzed included subjects with an observed ALT at 24 months.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 36 | 21
U/L | -3.7 (10) | 43.7 (239.5)

5. Secondary Outcome: Aspartate Aminotransferase (AST) Change From Baseline
Description: Liver function laboratory parameter
Time Frame: Baseline and 24 months
Population: Full analysis set, the # of subject analyzed included subjects with an observed AST at 24 months.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 35 | 21
U/L | -4.0 (8.5) | 31.4 (161.8)

6. Secondary Outcome: Caspase 3/7 Change From Baseline
Description: Mechanistic biomarker of liver function
Time Frame: Baseline and 24 months
Population: Full analysis set, the # of subject analyzed included subjects with an observed Caspase 3/7 at 24 months.
Measure: Mean (Standard Deviation); unit: Raw RLU
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 32 | 19
Raw RLU | -296.1 (830.3) | 2081.2 (10116.4)

7. Secondary Outcome: cCK18/M30 Change From Baseline
Description: Mechanistic biomarker of liver function.
Time Frame: Baseline and 24 months
Population: Full analysis set, the # of subject analyzed included subjects with an observed cCK18/M30 at 24 months.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 31 | 18
U/L | -104.7 (193.2) | -66.1 (176.9)

8. Secondary Outcome: flCK18/M65 Change From Baseline
Description: Mechanistic biomarker of liver function
Time Frame: Baseline and 24 months
Population: Full analysis set, the # of subject analyzed included subjects with an observed flCK18/M65 at 24 months.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 32 | 18
U/L | -70.2 (189.0) | -98.6 (311.7)

9. Secondary Outcome: Ishak Modification of Knodell Histological Activity Index - Interface Hepatitis
Description: The Ishak modification of Knodell histological activity index was determined by liver biopsy.
  Interface hepatitis
  * 0 = None
  * 1 = Mild (local, few portal areas)
  * 2 = Mild/moderate (focal, most portal areas)
  * 3 = Moderate (continuous around <50% of tracts or septa)
  * 4 = Severe (continuous around >50% of tracts or septa)
Time Frame: 24 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 41 | 23
Participants
  Interface Hepatitis Score of 0 | 6 | 5
  Interface Hepatitis Score of 1 | 14 | 4
  Interface Hepatitis Score of 2 | 8 | 6
  Interface Hepatitis Score of 3 | 3 | 1
  Interface Hepatitis Score of 4 | 1 | 3
  Missing Interface Hepatitis Score | 9 | 4

10. Secondary Outcome: Ishak Modification of Knodell Histological Index - Confluent Necrosis
Description: The Ishak modification of Knodell histological activity index will be determined by liver biopsy. The four items and their categorizations scores include:
  • confluent necrosis
  * 0 = None
  * 1 = Focal confluent necrosis
  * 2 = Zone 3 necrosis in some areas
  * 3 = Zone 3 necrosis in most areas
  * 4 = Zone 3 necrosis + occasional portal-central bridging
  * 5 = Zone 3 necrosis + multiple portal-central bridging
  * 6 = Panacinar or multiacinar necrosis
Time Frame: 24 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 41 | 23
Participants
  Confluent necrosis score of 0 | 32 | 19
  Missing confluent necrosis score | 9 | 4

11. Secondary Outcome: Ishak Modification of Knodell Histological Index - Parenchymal Injury
Description: The Ishak modification of Knodell histological activity index will be determined by liver biopsy.
  • parenchymal injury (focal lytic necrosis, apoptosis and focal inflammation)
  * 0 = None
  * 1 = One focus or less per 10× objective
  * 2 = Two to four foci per 10× objective
  * 3 = Five to ten foci per 10× objective
  * 4 = More than ten foci per 10× objective
Time Frame: 24 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 41 | 23
Participants
  Parenchymal Injury Score of 0 | 1 | 2
  Parenchymal Injury Score of 1 | 22 | 9
  Parenchymal Injury Score of 2 | 5 | 7
  Parenchymal Injury Score of 3 | 4 | 1
  Missing Parenchymal Injury Score | 9 | 4

12. Secondary Outcome: Ishak Modification of Knodell Histological Index - Portal Inflammation
Description: Portal inflammation
  * 0 = None
  * 1 = Mild, some or all portal areas
  * 2 = Moderate, some or all portal areas
  * 3 = Moderate/marked, all portal areas
  * 4 = Marked, all portal areas
Time Frame: 24 months
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | IDN-6556 | Placebo
Number analyzed (Participants) | 41 | 23
Participants
  Portal Inflammation Score of 1 | 11 | 4
  Portal Inflammation Score of 2 | 19 | 8
  Portal Inflammation Score of 3 | 2 | 6
  Portal Inflammation Score of 4 | 0 | 1
  Missing Portal Inflammation Score | 9 | 4

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from the first day of study drug administration until the subject's last study follow-up visit. All treatment emergent adverse events were collected up to the subsequent follow-up visit of the month 24 month visit.
Arm/Group | IDN-6556 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 1/23
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/23
Other Adverse Events (participants affected / at risk) | 37/41 | 20/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDN-6556 (N=41) | Placebo (N=23)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDN-6556 (N=41) | Placebo (N=23)
Diarrhea (Gastrointestinal disorders) | 9 (10) | 5 (6)
Hypertension (Vascular disorders) | 6 (7) | 4 (9)
Nausea (Gastrointestinal disorders) | 7 (10) | 5 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (10) | 2 (7)
Fatigue (General disorders) | 8 (8) | 6 (7)
Abdominal pain (Gastrointestinal disorders) | 4 (6) | 2 (2)

LIMITATIONS AND CAVEATS:
The broad range of fibrosis stages included in the study and the high placebo response rates especially in the F2 and F6 fibrosis stages impacted the primary endpoint of improvement in fibrosis score from baseline.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right to publish the results before the PI.

DOCUMENTS (2):
  • Study Protocol (2015-08-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT02138253/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-18): https://cdn.clinicaltrials.gov/large-docs/53/NCT02138253/SAP_001.pdf